CLINICAL TRIAL: NCT01522820
Title: A Phase I Clinical Trial of mTOR Inhibition With Rapamycin for Enhancing Intranodal Dendritic Cell Vaccine Induced Anti-tumor Immunity in Patients With NY-ESO-1 Expressing Solid Tumors
Brief Title: Vaccine Therapy With or Without Sirolimus in Treating Patients With NY-ESO-1 Expressing Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 191511; NCI-2011-03568 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 071614; I 191511 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH); R01CA158318 (NIH)
Record Dates: First submitted 2012-01-25; First posted 2012-02-01 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Anaplastic Astrocytoma; Anaplastic Oligoastrocytoma; Anaplastic Oligodendroglioma; Estrogen Receptor Negative; Estrogen Receptor Positive; Glioblastoma; Hormone-Resistant Prostate Cancer; Metastatic Prostate Carcinoma; Metastatic Renal Cell Cancer; Recurrent Adult Brain Neoplasm; Recurrent Bladder Carcinoma; Recurrent Breast Carcinoma; Recurrent Colorectal Carcinoma; Recurrent Esophageal Carcinoma; Recurrent Gastric Carcinoma; Recurrent Hepatocellular Carcinoma; Recurrent Lung Carcinoma; Recurrent Melanoma; Recurrent Ovarian Carcinoma; Recurrent Prostate Carcinoma; Recurrent Renal Cell Carcinoma; Recurrent Uterine Corpus Carcinoma; Resectable Hepatocellular Carcinoma; Sarcoma; Stage IA Breast Cancer; Stage IA Ovarian Cancer; Stage IA Uterine Corpus Cancer; Stage IB Breast Cancer; Stage IB Ovarian Cancer; Stage IB Uterine Corpus Cancer; Stage IC Ovarian Cancer; Stage II Uterine Corpus Cancer; Stage IIA Breast Cancer; Stage IIA Lung Carcinoma; Stage IIA Ovarian Cancer; Stage IIB Breast Cancer; Stage IIB Esophageal Cancer; Stage IIB Lung Carcinoma; Stage IIB Ovarian Cancer; Stage IIB Skin Melanoma; Stage IIC Ovarian Cancer; Stage IIC Skin Melanoma; Stage IIIA Breast Cancer; Stage IIIA Esophageal Cancer; Stage IIIA Lung Carcinoma; Stage IIIA Ovarian Cancer; Stage IIIA Skin Melanoma; Stage IIIA Uterine Corpus Cancer; Stage IIIB Breast Cancer; Stage IIIB Esophageal Cancer; Stage IIIB Ovarian Cancer; Stage IIIB Skin Melanoma; Stage IIIB Uterine Corpus Cancer; Stage IIIC Breast Cancer; Stage IIIC Esophageal Cancer; Stage IIIC Ovarian Cancer; Stage IIIC Skin Melanoma; Stage IIIC Uterine Corpus Cancer; Stage IV Bladder Urothelial Carcinoma; Stage IV Esophageal Cancer; Stage IV Ovarian Cancer; Stage IV Prostate Cancer; Stage IV Skin Melanoma; Stage IVA Uterine Corpus Cancer; Stage IVB Uterine Corpus Cancer
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Prostatic Neoplasms; Carcinoma, Renal Cell; Brain Neoplasms; Urinary Bladder Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Carcinoma, Hepatocellular; Lung Neoplasms; Melanoma; Ovarian Neoplasms; Sarcoma | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1a (vaccine therapy) (Experimental): Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401 protein vaccine intranodally on days 1, 29, 57, and 113.
  Interventions: Biological: DEC-205/NY-ESO-1 Fusion Protein CDX-1401; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Cohort 1b (vaccine therapy and immunotherapy) (Experimental): Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401 as in Cohort 1a and sirolimus PO or PEG on days 1-14, 29-42, and 57-70.
  Interventions: Biological: DEC-205/NY-ESO-1 Fusion Protein CDX-1401; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sirolimus
- Cohort 1c (vaccine therapy and immunotherapy) (Experimental): Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401 vaccine as in Cohort 1a and sirolimus PO or PEG on days 15-28, 43-56, and 71-84.
  Interventions: Biological: DEC-205/NY-ESO-1 Fusion Protein CDX-1401; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sirolimus
- Cohort 1d (vaccine therapy and immunotherapy) (Experimental): Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401 as in Cohort 1a and sirolimus PO or PEG on days 1-84.
  Interventions: Biological: DEC-205/NY-ESO-1 Fusion Protein CDX-1401; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sirolimus
- Cohort 2 (vaccine therapy with or without immunotherapy) (Experimental): Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401 as in the Cohort (1a-1d) that is determined to be safe and produces optimal immunological effects and sirolimus PO on days 1-14 as in Cohort 1b dose.
  Interventions: Biological: DEC-205/NY-ESO-1 Fusion Protein CDX-1401; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sirolimus

INTERVENTIONS:
Biological: DEC-205/NY-ESO-1 Fusion Protein CDX-1401 — Given intranodally
  Other Names: CDX-1401
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Sirolimus — Given PO or PEG
  Other Names: AY 22989; RAPA; Rapamune; RAPAMYCIN; SILA 9268A; WY-090217
  Arms: Cohort 1b (vaccine therapy and immunotherapy); Cohort 1c (vaccine therapy and immunotherapy); Cohort 1d (vaccine therapy and immunotherapy); Cohort 2 (vaccine therapy with or without immunotherapy)

SUMMARY:
This phase I trial studies the side effects and best schedule of vaccine therapy with or without sirolimus in treating patients with cancer-testis antigen (NY-ESO-1) expressing solid tumors. Biological therapies, such as sirolimus, may stimulate the immune system in different ways and stop tumor cells from growing. Vaccines made from a person's white blood cells mixed with tumor proteins may help the body build an effective immune response to kill tumor cells that express NY-ESO-1. Infusing the vaccine directly into a lymph node may cause a stronger immune response and kill more tumor cells. It is not yet known whether vaccine therapy works better when given with or without sirolimus in treating solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety of DC205-NY-ESO-1 vaccine (DEC-205/NY-ESO-1 fusion protein CDX-1401) with and without sirolimus. Toxicity as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OBJECTIVES:

I. Assess the NY-ESO-1 specific cellular and humoral immunity:

* Peripheral blood NY-ESO-1 specific cluster of differentiation (CD)8+ and CD4+ T-cells.
* Peripheral blood NY-ESO-1 specific antibodies.
* Peripheral blood frequency of CD4+CD25+forkhead box P3 (FOXP3)+ regulatory T-cells.

TERTIARY OBJECTIVES:

I. Explore time to disease progression.

OUTLINE:

Patients undergo standard collection of peripheral white blood cells via leukapheresis over 90-240 minutes for vaccine preparation. Patients are assigned sequentially to Cohorts 1a-1d.

COHORT 1a: Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401 intranodally on days 1, 29, 57, and 113.

COHORT 1b: Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401 as in Cohort 1a and sirolimus orally (PO) on days 1-14, 29-42, and 57-70.

COHORT 1c: Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401 as in Cohort 1a and sirolimus PO or percutaneous endoscopic gastrostomy (PEG) tube on days 15-28, 43-56, and 71-84.

COHORT 1d: Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401 as in Cohort 1a and sirolimus PO or PEG on days 1-84.

COHORT 2: Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401 as in the Cohort (1a-1d) that is determined to be safe and produces optimal immunological effects and sirolimus PO on days 1-14 as in Cohort 1b dose.

After completion of study treatment, patients are followed up at 6 weeks, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any solid tumors at high risk of recurrence or with minimal residual disease; there may or may not be measurable or symptomatic disease (i.e., patients with bladder, brain, breast, esophageal, gastrointestinal, hepatocellular, kidney, lungs, melanoma, ovarian, prostate, sarcomas, and uterine)
* Cancer types:

  * Prostate cancer: patients with metastatic, castrate refractory prostate cancer; the use of luteinizing hormone-releasing hormone (LHRH) agonist is allowed
  * Kidney cancer: patients with metastatic kidney cancer; prior therapies with cytokines, vascular endothelial growth factor (VEGF) and mechanistic target of rapamycin (serine/threonine kinase) (mTOR) inhibitors are allowed
  * Bladder cancer: patients with metastatic urothelial carcinoma; prior cisplatin-based therapies are allowed
  * Ovarian cancer: eligible patients may have asymptomatic residual measurable disease on physical examination and/or computed tomography (CT) scan, and/or may have an elevated cancer antigen (CA)-125; or may be in complete clinical remission after treatment for primary or recurrent disease
  * Brain tumors: histologic proof of one of the following: glioblastoma multiforme, anaplastic astrocytoma, anaplastic oligodendroglioma or anaplastic mixed glioma or anaplastic oligoastrocytoma; patients who have had recent cranial surgery are eligible for inclusion, but the vaccine may not be administered prior to postoperative day 14
  * Uterine cancer: patients with advanced (stages II-IV) or recurrent disease who have completed standard therapy, currently no evidence of disease (NED) or with minimal residual disease; patients with stage I uterine serous carcinomas or sarcomas are also eligible after completion of standard therapy
  * Breast cancer: patients can enter study after completion of all chemotherapy (including trastuzumab), radiation, and breast/axillary surgery; patients may participate while on endocrine therapy; stages I-III patients with the following characteristics:

    * Estrogen-receptor (ER) negative with positive lymph nodes; ER negative with negative nodes if tumor > 2 cm; ER positive with positive lymph nodes; and ER positive with negative lymph nodes and tumor > 5 cm
  * Sarcomas: patients with sarcomas of any site, who have completed standard therapy, and are in remission, or have minimal disease burden
  * Lungs: resected patients with hilar or ipsilateral mediastinal nodal disease (i.e., a subset of patients with stage II and IIIA disease); and patients with residual disease on imaging after definitive radiation or chemoradiation therapy
  * Esophageal: resected patients with any nodal (i.e., thoracic or abdominal) disease; and patients with residual disease on imaging after definitive chemoradiation therapy
  * Melanoma: stage IIB, stage IIC, and stage III who have completed planned definitive therapy for their disease including radiotherapy and/or interferon; patients declining interferon or with contra-indications to interferon will also be eligible provided they meet requisite criteria for this study (i.e., non-measurable disease); stage IV melanoma of M1a sub-type only, who are not candidates for additional therapy of curative potential (i.e., small volume disease; may be measurable or evaluable); and stage IV melanoma, NED, status post (s/p) complete resection of known sites of disease (i.e., non-measurable disease)
  * Hepatocellular carcinoma (HCC): patients who have been treated with surgical resection for HCC; and following chemoembolization as adjuvant therapy for HCC
  * Gastrointestinal: patients who have completed standard therapies for gastric and colorectal cancers, and deemed to be at high-risk of relapse
* Any human leukocyte antigen (HLA) type; historic HLA typing is permitted
* Tumor expression of NY-ESO-1 or LAGE-1 by immunohistochemistry (IHC) and/or reverse transcription polymerase chain reaction (RTPCR)
* Life expectancy > 6 months
* Absolute neutrophil count (ANC) >= 1,000/uL
* Platelets (PLT) >= 75,000/uL
* Hemoglobin (Hgb) >= 8 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Serum aspartate aminotransferase (serum glutamic oxaloacetic transaminase [SGOT]/aspartate aminotransferase [AST]) or serum alanine aminotransferase (serum glutamate pyruvate transaminase [SGPT]/alanine aminotransferase [ALT]) =< 3 x ULN
* Serum creatinine =< 2 x ULN
* Prothrombin time (PT)/international normalized ratio (INR) =< 1.5 x ULN; patients receiving anticoagulation therapy, PT/INR =< 3
* Pulmonary function tests: forced expiratory volume in one second (FEV1) > 50% and diffusion capacity of the lungs for carbon monoxide (DLCO) > 50%
* Pulse oximetry: oxygen (O2) saturation >= 90% on room air
* Electrocardiogram, showing no clinical significant or acute abnormality
* Have been informed of other treatment options
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Patients of child-bearing potential must agree to use acceptable contraceptive methods (e.g., double barrier) during treatment

Exclusion Criteria:

* Metastatic disease to the central nervous system for which other therapeutic options, including radiotherapy, may be available
* Other serious illnesses (e.g., serious infections requiring antibiotics, bleeding disorders)
* History of severe autoimmune disorders requiring use of steroids or other immunosuppressives
* Concomitant systemic treatment with corticosteroids, anti-histamine or non-steroidal anti-inflammatory drugs, aspirin > 325 mg; specific cyclooxygenase (COX)-2 inhibitors are permitted
* Chemotherapy, radiation therapy, or immunotherapy within 4 weeks prior to first dosing of study agent (6 weeks for nitrosoureas); concomitant hormonal therapies for breast and prostate cancers are allowed
* Clinically significant heart disease (New York Heart Association [NYHA] class III or IV) within 6 months
* Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study
* Lack of availability of a patient for immunological and clinical follow-up assessment
* Known pulmonary hypertension
* Known hypersensitivity to sirolimus
* Evidence of current drug or alcohol abuse or psychiatric impairment, which in the investigator's opinion will prevent completion of the protocol therapy or follow-up
* Pregnant or nursing female patients
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the patient an unsuitable candidate to receive study drug; (i.e., any significant medical illness or abnormal laboratory finding that would, in the investigator's judgment, increase the subject's risk by participating in this study)
* Received an investigational agent within 30 days prior to enrollment
* Known hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events in patients receiving the DEC-205/NY-ESO-1 fusion protein CDX-1401 with and without sirolimus, as evaluated according to the NCI CTCAE scale version 4.0 | Up to 12 months post-treatment
  The safe schedule of the combinatorial regimen is established at the dose before 2/6 patients experience dose-limiting toxicity. Estimated using a one-sided, 95%, exact binomial confidence interval (Clopper-Pearson).

SECONDARY OUTCOMES:
NY-ESO-1 specific cellular immunity | Up to 12 months post-treatment
  Analyzed via an analysis-of-covariance (ANCOVA) model with post-treatment levels modeled as a function pretreatment levels and main effects corresponding to the 3 + 3 design.
NY-ESO-1 specific humoral immunity | Up to 12 months post-treatment
  ANCOVA model with post-treatment levels modeled as a function pretreatment levels and main effects corresponding to the 3 + 3 design.

OTHER OUTCOMES:
Time to disease progression | Up to 12 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kunle Odunsi, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] Withers HG, Matsuzaki J, Long M, Rosario SR, Chodon T, Tsuji T, Koya R, Yan L, Wang J, Keler T, Lele SB, Zsiros E, Lugade A, Hutson A, Blank S, Bhardwaj N, Shrikant P, Liu S, Odunsi K. mTOR inhibition modulates vaccine-induced immune responses to generate memory T cells in patients with solid tumors. J Immunother Cancer. 2025 Mar 25;13(3):e010408. doi: 10.1136/jitc-2024-010408. PMID 40132910